CLINICAL TRIAL: NCT01844908
Title: Can Electroacupuncture Prevent Prolonged Ileus After Laparoscopic Surgery for Mid and Low Rectal Cancer? A Prospective Study With Matched Historical Controls
Brief Title: Electroacupuncture for Postoperative Ileus After Laparoscopic Rectal Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2013.032
Record Dates: First submitted 2013-04-24; First posted 2013-05-03 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electroacupuncture (Experimental)
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture

SUMMARY:
Postoperative ileus remains a significant medical problem after colorectal surgery that adversely influences patients' recovery. The investigators previous study demonstrated that electroacupuncture (EA) at Zusanli, Sanyinjiao, Hegu, and Zhigou reduces the duration of postoperative ileus and hospital stay after laparoscopic resection of colonic and upper rectal cancer. Patients with mid/low rectal cancer undergoing laparoscopic total mesorectal excision (TME) or abdominoperineal resection (APR) were excluded. However, these complex cases are more likely to develop prolonged ileus and morbidity after surgery, and it is uncertain whether EA will be beneficial to them. The investigators therefore propose to conduct a prospective cohort study to evaluate the efficacy of EA in preventing prolonged ileus after laparoscopic surgery for mid/low rectal cancer. Fifty consecutive patients with mid/low rectal cancer undergoing laparoscopic TME or APR without the need of conversion will be recruited. All patients will undergo 1 session (20 minutes) of EA daily from postoperative day 1 till day 4. These patients will be compared with a matched historical control group (1:2) who underwent laparoscopic TME or APR without EA. The primary outcome is the incidence of prolonged ileus, which is defined as the inability to tolerate fluid diet by 4 days after surgery, associated with the need for nasogastric decompression and/or parenteral nutrition support. Secondary outcomes include time to defecation and duration of hospital stay. Results of this study will help clarify the efficacy of EA in preventing prolonged ileus after laparoscopic rectal surgery, and may provide the basis for planning a larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients (aged between 18 and 80) with mid/low rectal cancer undergoing laparoscopic TME or APR without the need of conversion
* Patients with American Society of Anesthesiologists grading I-III
* Informed consent available

Exclusion Criteria:

* Patients undergoing simultaneous laparoscopic resection of rectal cancer and other coexisting intraabdominal diseases
* Patients undergoing laparoscopic resection of rectal cancer with en-bloc resection of surrounding organs
* Patients who developed intraoperative problems or complications (e.g. bleeding, tumor perforation) that required conversion
* Patients with intestinal obstruction
* Patients with previous history of abdominal surgery
* Patients with evidence of peritoneal carcinomatosis
* Patients who are expected to receive epidural anesthesia or analgesia
* Patients with cardiac pacemaker
* Patients who are pregnant
* Patients who are allergic to acupuncture needles

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of prolonged ileus | Up to 1 month
  Defined as the inability to tolerate fluid diet by 4 days after surgery, associated with the need for nasogastric decompression and/or parenteral nutrition support.

SECONDARY OUTCOMES:
Time of first passing flatus reported by the patients | Up to 1 month
Time to first defecation | Up to 1 month
Time that the patients tolerated solid diet | Up to 1 month
Duration of hospital stay | Up to 1 month
Pain scores on visual analog scale | Up to 3 days
  From 0 which implies no pain at all, to 10 which implies the worst pain imaginable
Postoperative analgesic requirement | Up to 1 month
Overall complication rate | Up to 1 month
30-day mortality rate | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong SAR, China